CLINICAL TRIAL: NCT02920216
Title: Pilot Study of Evaluation of the Interest of Fluorescence in Salvage Surgery for Recurrence of Head and Neck Cancer in Irradiated Area
Brief Title: Interest of Fluorescence in Salvage Surgery for Recurrence of Head and Neck Cancer in Irradiated Area
Acronym: SALVADS-Fluo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A00014-47
Record Dates: First submitted 2016-09-21; First posted 2016-09-30 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Neoplasms; Recurrence; Indocyanine Green; Salvage surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eligible patient for a salvage surgery (Experimental)
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — intravenous injection of Indocyanine Green (0,25mg/kg) before surgery.

SUMMARY:
Treatment of Head and Neck Squamous cell carcinoma often combines chemoradiotherapy when organ has to be preserved or when surgery is not indicated. The loco-regional failure is about 30%. Then salvage surgery is the only chance for patients to survive but the overall survival rate is only 29% at 24 months. This prognostic is bad because of poor local control which is non-optimized by a complementary radiotherapy and negative exeresis margins.

Currently, there is no intraoperative technique to better visualize the tumor limits in real time. With fluorescence techniques, an accurate mapping of tumor extension can be considered. Recently, Atallah et al. (2015) demonstrated the use of fluorescence during a head and neck surgery in mice, as a tool allowing for better surgical margins. Digonnet et al (2015) found a tumor fragment after an injection of indocyanine green (ICG) intravenously in salvage surgery for patient with head and neck cancer.

The ability of ICG to detect a surgical margin positive intraoperatively has never be evaluated in irradiated area.

The aim of this pilot study is to evaluate the interest of fluorescence in salvage surgery for recurrence of head and neck cancer in irradiated area.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Head and Neck Squamous Cell Carcinoma confirmed by biopsy
* Non metastatic disease
* Resectable tumour
* Locoregional recurrence or new localization in pre irradiated territory at a dose ≥ 50 Gy with or without chemotherapy
* Haematological constants, liver function and kidney function adapted in the 15 days before inclusion:

  * Haemoglobin ≥ 9 g / dL
  * Polymorphonuclear neutrophils ≥ 1.5 x 10 9
  * Platelet ≥ 100 x 109 / L
  * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * ALT and AST <3 times ULN
  * Alkaline phosphatase ≤ 2.5 times ULN
  * Serum creatinine <110 mmol / L or creatinine clearance> 55 ml / min (method of Cockcroft)
  * Absence of proteinuria
* WHO 0 or 1
* Signed informed consent form
* Patient affiliated to the social security system.

Exclusion Criteria:

* Patient considered as non eligible for a salvage surgery
* Metastatic disease
* Hypersensitivity to indocyanine green or allergy to seafood or reaction to iodinated contrast agents
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of indocyanine green labeling in Irradiated Area | 1 day
  The indocyanine green labeling in irradiated areas will be compared to the histological result on the surgical specimen.

SECONDARY OUTCOMES:
Sensitivity of indocyanine green labeling on surgical margins | 1 day
  The indocyanine green labeling on surgical margins will be compared to the surgical margins histological result

CONTACTS AND LOCATIONS:
Overall Officials: CORTESE Sophie, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cortese S, Kerrien E, Yakavets I, Meilender R, Mastronicola R, Renard S, Leroux A, Bezdetnaya L, Dolivet G. ICG-induced NIR fluorescence mapping in patients with head & neck tumors after the previous radiotherapy. Photodiagnosis Photodyn Ther. 2020 Sep;31:101838. doi: 10.1016/j.pdpdt.2020.101838. Epub 2020 May 30. PMID 32479902